CLINICAL TRIAL: NCT05556551
Title: Clinical Performance of Lithium Disilicate Versus Hybrid Resin Ceramic for Inlay and Onlay Restoration After 3 Years Follow up
Brief Title: Comparing Between Two Different Restoration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 7755100
Record Dates: First submitted 2022-09-05; First posted 2022-09-27 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2019-09

CONDITIONS: Dental Restoration Failure

STUDY DESIGN:
Intervention Model Description: Two different restorations in patient mouth
Who Masked: Participant
Masking Description: Different restoration inserted in the patient mouth
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hybrid resin ceramic restoration (Other): Dental restoration
  Interventions: Other: Hybrid resin Ceramic restoration
- Full ceramic restoration (Other): Dental restoration
  Interventions: Other: Full Ceramic restoration

INTERVENTIONS:
Other: Full Ceramic restoration — Two different dental restoration inserted in patient mouth ( split mouth)
  Arms: Full ceramic restoration
Other: Hybrid resin Ceramic restoration — Hybrid resin Ceramic restoration
  Arms: Hybrid resin ceramic restoration

SUMMARY:
Clinical performance of two different ceramic restoration in patient mouth after 3 years follow up

DETAILED DESCRIPTION:
Comparing two different dental restoration in patient mouth after 3 years follow up by using USPHS criteria

ELIGIBILITY:
Inclusion Criteria:

* good oral hygiene

Exclusion Criteria:

* bad oral hygiene

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2019-05-20 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of two different restoration | 3 years
  Using (USPHS) criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Amr hany hassan, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No
Evaluation of two different restoration after 3 years follow up

REFERENCES:
- [Background] Rubinstein MH. A new granulation method for compressed tablets [proceedings]. J Pharm Pharmacol. 1976 Dec;28 Suppl:67P. No abstract available. PMID 12345